CLINICAL TRIAL: NCT02354859
Title: A Phase 2, Multi-Center, Randomized, Placebo-Controlled Study of IV Gallium Nitrate in Patients With Cystic Fibrosis (IGNITE Study)
Brief Title: A Phase 2 IV Gallium Study for Patients With Cystic Fibrosis (IGNITE Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Chris Goss, Professor, Medicine/Pulmonary & Critical Care Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002609; 2R01FD003704-03A1 (FDA)
Record Dates: First submitted 2014-07-30; First posted 2015-02-03 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Gallium Nitrate; IV Gallium; Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — gallium nitrate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 day of infusion of gallium nitrate (Active Comparator): Gallium nitrate will be infused continuously over 5 days at 200 mg/m2/day. Study drug will be administered via a peripheral IV catheter, a peripherally inserted central catheter (PICC) line, midline catheter, or a chronic indwelling vascular access device () using an ambulatory infusion pump infused over 24 hours for 5 sequential days.
  Interventions: Drug: Gallium nitrate
- 5 day of infusion of normal saline (Placebo Comparator): Placebo with be dispensed as 1,000 milliliters of 0.9% sodium chloride to match the reconstitution volume of the IV Ga
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Gallium nitrate — Study subjects will receive an infusion of either placebo or gallium nitrate.
  Other Names: Ga, GaN3O9
  Arms: 5 day of infusion of gallium nitrate
Drug: Normal Saline — Study subjects will receive an infusion of either placebo (normal saline) or gallium nitrate.
  Other Names: Sodium Chloride, NS
  Arms: 5 day of infusion of normal saline

SUMMARY:
The purpose of this study is to assess the efficacy of IV gallium to improve pulmonary function as measured by a 5% or greater relative improvement in forced expiratory volume in one second (FEV1) from baseline to Day 28.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
This is a phase 2, multi-center, randomized, placebo-controlled trial in adults with CF chronically infected with P. aeruginosa. The study will evaluate the safety and clinical efficacy of a five day infusion of IV gallium nitrate (IV gallium). The purpose of this study is to assess the efficacy of IV gallium to improve pulmonary function as measured by a 5% or greater relative improvement in forced expiratory volume in one second (FEV1) from baseline to Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age at Screening
* Documented chronic colonization with P. aeruginosa defined as dentification in two sputum or oropharyngeal cultures within the year prior to Day 1
* Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

  1. sweat chloride ≥ 60 mEq/liter by quantitative pilocarpine iontophoresis test (QPIT)
  2. two well-characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
  3. Abnormal nasal potential difference (NPD; change in NPD in response to a low chloride solution and isoproteronol of less than -5 mV)
* FEV1 ≥ 25 % of predicted value at Screening
* Able to expectorate sputum
* Serum liver function tests ≤ 2.5 x upper limit of normal at Screening
* Serum urea nitrogen (BUN) ≤ 1.5 x upper limit of normal at Screening
* Serum creatinine ≤ 2.0 mg/dl and ≤ 1.5 x upper limit of normal at Screening
* Hemoglobin ≥ 9 g/dl, platelets ≥ 100,000/mm3, and white blood cells (WBC)

  ≥ 4,500/mm3 at Screening
* Ionized calcium ≥ lower limit of normal at Screening
* Written informed consent obtained from subject or subject's legal representative
* Able to communicate with the Investigator and comply with the requirements of the protocol
* If female and of childbearing potential, must have a negative pregnancy test on Day 1 prior to receiving study drug
* If female and of childbearing potential, is willing to use adequate contraception for the duration of the study through Visit 5, as determined by the investigator
* If male and able to father a child, is willing to use adequate contraception for the duration of the study through Visit 5, as determined by the investigator
* Clinically stable with no significant changes in health status within 14 days prior to Day 1

Exclusion criteria:

* Use of inhaled antibiotics within seven days prior to Day 1
* Unable or unwilling to withhold use of chronic inhaled antibiotics through Day 28
* Use of intravenous, inhaled, or oral antibiotics for an acute indication within 14 days prior to Day 1
* Use of bisphosphonates within seven days prior to Day 1
* History of osteoporosis (defined as the most recent dexa scan with a T-score ≤ -2.5 with the dexa scan performed within the five years prior to Screening)
* Lactating female
* Known sensitivity to gallium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Goss, MD, Principal Investigator — University of Washington
Locations (23):
- United States (23):
  - AL Adult Birmingham / The Children's Hospital Atlanta, Birmingham, Alabama
  - UC San Diego Medical Center, La Jolla, California
  - Denver Adult / National Jewish Health, Denver, Colorado
  - Shands Hospital, Gainesville, Florida
  - Jackson Memorial Hospital; University of Miami Hospital; University of Miami Hospital and Clinics, Miami, Florida
  - Atlanta Emory Adult / Emory University Hospital, Atlanta, Georgia
  - Chicago Northwestern Adult / Northwestern Memorial Hospital, Chicago, Illinois
  - Iowa City University of Iowa Adult / University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Lexington, KY Adult / University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Portland, ME Adult, Portland, Maine
  - Baltimore Hopkins Adult / John Hopkins Hospital, Baltimore, Maryland
  - Boston CHB Adult / Boston Children's Hospital (BCH), Boston, Massachusetts
  - Minneapolis CC and Adult / University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Omaha Adult / The Nebraska Medical Center, Omaha, Nebraska
  - Lebanon, NH Dartmouth-Hitchcock CC and Adult / Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cleveland CC and Peds, Hospital of Cleveland, Cleveland, Ohio
  - Columbus CC and Peds / Nationwide Children's Hospital, Columbus, Ohio
  - Toledo, OH CC and Peds / The Toledo Hospital; Toledo Children's Hospital, Toledo, Ohio
  - Oklahoma City Adult / Presbyterian Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - Pittsburgh Adult, Children's Hospital of Pittsburgh UPMC, Pittsburgh, Pennsylvania
  - SC CC and Adult Charleston / MUSC, Charleston, South Carolina
  - Salt Lake City Adult, Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - Seattle UW Adult / University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Once the study is complete and the primary paper is published, de-identified data will be available from the Cystic Fibrosis Therapeutics Development Network Coordinating Center upon approval of a formal data request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Gallium: Gallium nitrate will be infused continuously over 5 days at 200 mg/m2/day. Study drug will be administered via a peripheral IV catheter, a peripherally inserted central catheter (PICC) line, midline catheter, or a chronic indwelling vascular access device () using an ambulatory infusion pump infused over 24 hours for 5 sequential days.
  Gallium nitrate: Study subjects will receive an infusion of either placebo or gallium nitrate.
- Placebo: Placebo with be dispensed as 1,000 milliliters of 0.9% sodium chloride to match the reconstitution volume of the IV Ga
  Normal Saline: Study subjects will receive an infusion of either placebo (normal saline) or gallium nitrate.
Period: Overall Study
Arm/Group | Gallium | Placebo
Started (Treated, defined as randomized and started on study drug (IV gallium or placebo)) | 60 | 59
Completed (Completed last study visit (Day 56)) | 60 | 57
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gallium | Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (10.25) | 33.8 (9.62) | 32.8 (9.96)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution: Between 18 and 30 years | 30 | 23 | 53
  Age Distribution: >= 30 years | 30 | 36 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 29 | 35 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 58 | 58 | 116
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants] — Other refers to participants with either two known, non-F508 del CF mutations, or one known, non-F508 del CF mutation and one unidentified allele which has not been classified as a CF mutation. Unidentified refers to participants with 2 alleles that have not been classified as CF mutations.
  Participants
    Delta F508 Homozygous | 34 | 38 | 72
    Delta F508 Heterozygous | 21 | 18 | 39
    Other | 5 | 2 | 7
    Unidentified | 0 | 0 | 0
    Not Available | 0 | 1 | 1
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.0 (0.95) | 2.0 (0.79) | 2.0 (0.87)
FEV1 (% Predicted) Distribution [Count of Participants; unit: Participants] — FEV1 (% predicted) is calculated using the Hankinson reference equations.
  Participants
    < 50% | 28 | 29 | 57
    Between 50 and 70% | 15 | 12 | 27
    > 70% | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 5% or Greater Relative Change in FEV1 (Liters) From Baseline to Day 28
Description: Difference between treatment groups in the proportion of subjects with 5% or greater relative change in FEV1 (liters) from baseline to Day 28.
Time Frame: Baseline to Day 28
Population: Includes only treated participants with FEV1 measurements at Baseline and Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 60 | 56
Participants | 22 | 17
Statistical Analysis 1: Comparison: Gallium vs Placebo; Test type: Superiority; p = 0.811, Cochran-Mantel-Haenszel; Difference in Proportions = 5.9, 95% CI 2-sided [-11.2 to 22.4] — The estimate is adjusted for baseline FEV1 % predicted strata (<50% of predicted, between 50% and 70% of predicted, and >70% of predicted)

2. Secondary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Incidence is defined as the number and percentage of participants with at least one event over the 56 day follow-up period.
Time Frame: Day 1 to Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 60 | 59
Participants
  Incidence of AEs | 57 | 57
  Incidence of SAEs | 11 | 9
Statistical Analysis 1: Comparison: Gallium vs Placebo; Test type: Superiority; p = 0.807, Fisher Exact; Difference in Proportions-SAE inicidence = 3.1, 95% CI 2-sided [-10.6 to 16.6] — 95% confidence interval calculated using the Newcombe-Wilson method without continuity correction

3. Secondary Outcome: Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Rate is defined as the number of events per participant follow-up week.
Time Frame: Day 1 to Day 56
Measure: Number; unit: events per participant-week
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 60 | 59
events per participant-week
  Number of AEs per participant week | 0.84 | 1.03
  Number of SAEs per participant week | 0.02 | 0.03
Statistical Analysis 1: Comparison: Gallium vs Placebo; Rate Ratio for Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks of all participants (not per participant) in the trial was as follows: in the IV Gallium group was 486.86 and in the Placebo group was 473.57; Test type: Superiority; p = 0.002, Poisson Regression; Rate Ratio = 0.81, 95% CI 2-sided [0.71 to 0.93]
Statistical Analysis 2: Comparison: Gallium vs Placebo; Rate Ratio for Serious Adverse Events calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks in the IV Gallium group was 486.86 and in the Placebo group was 473.57; Test type: Superiority; p = 0.783, Poisson Regression; Rate Ratio = 0.89, 95% CI 2-sided [0.39 to 2.03]

4. Secondary Outcome: Relative Change in FEV1 (Liters) From Baseline to Day 56
Description: Difference between treatment groups in the relative change in FEV1 (liters) from Baseline to Day 56
Time Frame: Day 1 to Day 56
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 60 | 59
percentage change | 1.89 (16.99) | -0.05 (14.14)
Statistical Analysis 1: Comparison: Gallium vs Placebo; Test type: Superiority; p = 0.479, Mixed Models Analysis; Mean Difference (Final Values) = 2.05, 95% CI 2-sided [-3.66 to 7.77] — Analysis includes all data for relative change from baseline at Day 6, Day 14, Day 28, and Day 56. Mixed-effects repeated measures model includes terms for the baseline FEV1 (liters), treatment, visit and a visit-by-visit interaction

5. Secondary Outcome: Absolute Change in P. Aeruginosa Sputum Density (log10 (CFU)) From Baseline to Day 56
Description: Difference between treatment groups in the absolute change in P. aeruginosa sputum density (log10 (CFU)) from Baseline to Day 56 based on quantitative cultures.
Time Frame: Day 1 to Day 56
Population: Includes only participants with a positive P. aeruginosa (Pa) culture at Baseline.
Measure: Mean (Standard Error); unit: log10 (CFU)
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 47 | 45
log10 (CFU) | -1.06 (1.97) | -0.33 (1.52)
Statistical Analysis 1: Comparison: Gallium vs Placebo; Test type: Superiority; p = 0.054, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.49 to 0.01] — Analysis includes all data for relative change from baseline at Day 28 and Day 56. Mixed-effects repeated measures model includes terms for the baseline Pa density (log10 (CFU)), treatment, visit and a visit-by-visit interaction

6. Secondary Outcome: Absolute Change in Respiratory Symptoms, as Measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CFRSD-CRISS), From Baseline to Day 56
Description: Difference between treatment groups in the absolute change in respiratory symptoms, as measured by the the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CFRSD-CRISS), from Baseline to Day 56. The Cystic Fibrosis Respiratory Symptoms Daily Diary asks a participant to state the extent of their 8 respiratory symptoms : difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present 'a great deal' or 'extremely'. A summed score (range from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100, where the lowest scores indicate improvement of symptoms.
Time Frame: Day 1 to Day 56
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Gallium | Placebo
Number analyzed (Participants) | 60 | 59
score on a scale | 3.03 (13.66) | -0.98 (10.75)
Statistical Analysis 1: Comparison: Gallium vs Placebo; Test type: Superiority; p = 0.053, Mixed Models Analysis; Mean Difference (Final Values) = 4.23, 95% CI 2-sided [-0.06 to 8.53] — Analysis includes all data for relative change from baseline at Day 6, Day 14, Day 28, and Day 56. Mixed-effects repeated measures model includes terms for the baseline CFRSD-CRISS score, treatment, visit and a visit-by-visit interaction

ADVERSE EVENTS:
Time Frame: For Serious Adverse Events (SAEs): Informed consent to Day 56. For all Other (Not Including Serious) AEs: Start of study drug to final study visit (Day 56).
Arm/Group | Gallium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 11/60 | 9/59
Other Adverse Events (participants affected / at risk) | 53/60 | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gallium (N=60) | Placebo (N=59)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 3 (4)
Chills (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gallium (N=60) | Placebo (N=59)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 9 (13) | 11 (13)
Vomiting (Gastrointestinal disorders) | 4 (6) | 6 (6)
Asthenia (General disorders) | 6 (6) | 2 (2)
Chest discomfort (General disorders) | 12 (12) | 13 (15)
Chest pain (General disorders) | 5 (6) | 4 (5)
Chills (General disorders) | 0 (0) | 4 (4)
Fatigue (General disorders) | 19 (20) | 15 (16)
Pyrexia (General disorders) | 7 (7) | 14 (16)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Pulmonary function test decreased (Investigations) | 3 (3) | 3 (3)
Weight decreased (Investigations) | 4 (5) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 17 (20) | 23 (28)
Sinus headache (Nervous system disorders) | 2 (2) | 3 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (33) | 27 (34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 14 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 10 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (9)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (12)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 24 (30)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (11)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT02354859/SAP_000.pdf
  • Study Protocol (2014-08-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02354859/Prot_001.pdf